CLINICAL TRIAL: NCT06056128
Title: Confirmation of Accuracy of the Tool-in-lesion Technology (TiLT) of the Galaxy System With Integrated TOMO Technology in Human Subjects to Bronchoscopically Biopsy Small Peripheral Pulmonary Nodules: TiLT Study
Brief Title: Confirmation of Accuracy of the Tool-in-lesion Technology (TiLT) of the Galaxy System With Integrated TOMO Technology
Acronym: TiLT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Noah Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NOAH-002
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer; Nodes, Lung
Keywords: Lung cancer, robotic assisted bronchoscopy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Robotic assisted bronchoscopy (Experimental): Robotic assisted bronchoscopy procedures performed using the Galaxy System.
  Interventions: Device: Robotic assisted bronchoscopy

INTERVENTIONS:
Device: Robotic assisted bronchoscopy — Robotic assisted bronchoscopy of peripheral airways for the purpose of biopsying lung lesions

SUMMARY:
This study will evaluate the feasibility of performing robotic navigation of peripheral airways in human subjects for the purpose of biopsying peripheral lung lesions.

DETAILED DESCRIPTION:
Successful biopsy of peripheral pulmonary lesions continues to be a challenge due to a number of factors, one of which may be the ability to gain access to peripheral lesions due to the size and maneuverability of conventional bronchoscopes. In this study, investigators will evaluate the feasibility of the Galaxy System, which uses a built-in real-time navigation system called TiLT Technology, to both access and biopsy peripheral pulmonary lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Patients with a moderate to high risk of lung cancer based on clinical, demographic and radiologic information, determined by the treating physicians based on the site's standard of care
3. Peripheral pulmonary subsolid and solid nodules (PPNs) sized 1-3 cm measured as the largest dimension where all or the majority of the lesion is located in the periphery of the lung
4. Pre-procedural CT is conducted within 90 days of the bronchoscopy procedure
5. PPNs that are accessible bronchoscopically on planning CT reconstruction
6. Informed consent properly obtained per local regulations

Exclusion Criteria:

1. Known pregnancy or breastfeeding
2. Patients with pure ground-glass nodules on pre-procedural chest CT
3. Uncontrolled coagulopathy or bleeding disorders
4. Ongoing systemic infection
5. History of lobectomy or pneumonectomy
6. Patient is participating in another drug or device trial or participated in another drug or device trial in the last 30 days.
7. Moderate-to-severe hypoxia, hypoxemia, or hypercarbia per PI's discretion
8. Patients with pacemakers or defibrillators
9. Unsuitable for bronchoscopy procedure under general anaesthesia as agreed by the treating clinician and anaesthetist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Successful tool-in-lesion (defined as the tool within the lesion) as confirmed by CBCT. | During the procedure
  Successful navigation of the tool in lesion using the Galaxy System's TiLT technology will be confirmed using Cone Beam Computed Tomography (CBCT) prior to biopsies being performed.
Serious device or procedure related adverse events and device deficiencies during the bronchoscopy procedure and post-procedure | Up to 7 days post-procedure
  Number of patients with device or procedure related adverse events divided by number of patients who underwent the robotic bronchoscopy procedure.

SECONDARY OUTCOMES:
Diagnostic yield | Between 7 days and 6 months post-procedure
  Number of patients who are provided a definitive diagnosis based on the pathology report of the biopsied tissue.
Center strike as confirmed by CBCT | During the procedure
  Number of patients that the tool was confirmed to be in the center of the lesion prior to biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Calvin Ng, MD, Principal Investigator — Chinese University of Hong Kong, Prince of Wales Hospital
Locations (1):
- Chinese University of Hong Kong, Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No